CLINICAL TRIAL: NCT00949026
Title: Assessment of Systemically Administered Torisel Delivery to Brain Tumors by Intratumoral Microdialysis
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: No accrual
Sponsor: Emory University (Other)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Principal Investigator, Jeffrey James Olson, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00008256; WCI1388-07 (Other: Other)
Record Dates: First submitted 2009-07-29; First posted 2009-07-30 (Estimated); Last update posted 2013-11-21 (Estimated); Status verified 2013-11

CONDITIONS: Brain Neoplasms
Keywords: Brain Cancer; Brain Neoplasms, Malignant
MeSH Terms: conditions — Brain Neoplasms | interventions — temsirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental)
  Interventions: Drug: Temsirolimus (Torisel)

INTERVENTIONS:
Drug: Temsirolimus (Torisel) — Dose de-escalation dependent on microdialysis results
  Other Names: Torisel

SUMMARY:
The primary purpose of this study is to determine if it is effective to take samples of fluid from the patient's brain tumor with a microdialysis catheter for Torisel measurement. The investigators are also doing it to learn if it is safe to do so. The investigators will use these samples to measure how much Torisel reaches the patient's brain tumor. The use of the microdialysis catheter to collect brain fluid is an FDA approved method. This catheter is already being used in patients who have sustained severe brain trauma from head injuries. The catheter itself is smaller in size than the standard needle that will be used to take the patient's biopsy. To obtain additional information Torisel will also be measured at the same time in the patient's cerebral spinal fluid by taking it from a catheter placed in the patient's cerebral spinal fluid producing spaces in their brain and in their blood from a catheter in one of their vessels.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be at least 18 years of age.
2. Patients must have histologically confirmed supratentorial grade III or IV astrocytoma (anaplastic astrocytoma, anaplastic oligodendroglioma, glioblastoma multiforme) and require a stereotactic biopsy for confirmation of tumor progression or differentiation of tumor progression from treatment induced effects following radiation therapy ± chemotherapy. Patients with previous low-grade glioma who progressed after radiotherapy ± chemotherapy and are in need of a stereotactic biopsy to confirm the presence of a high-grade glioma, and this is accomplished at the time of biopsy, are eligible.
3. Patients must have a Karnofsky performance status ≥ 50% (i.e. the patient must be able to care for himself/herself with occasional help from others).
4. Patients must have had prior radiation therapy.
5. The patient is a candidate for temsirolimus as the next therapy for their tumor and the treating physician and the patient must be planning to continue temsirolimus chemotherapy after receiving the one dose required for this study.
6. Patients must have recovered from the toxicity of prior therapy. An interval of at least 3 months must have elapsed the since the completion of the most recent course of radiation therapy while at least 3 weeks must have elapsed since the completion of a non-nitrosourea containing chemotherapy regimen and at least six weeks since the completion of a nitrosourea containing chemotherapy regimen.
7. Patients must have adequate bone marrow function (defined as an absolute neutrophil count of >1500 cells/mm3 and platelet count >100,000 cells/mm3), liver function with Total bilirubin <2.0 mg/dl and SGOT <4 times upper limit of normal, and adequate renal function with serum creatinine ≤ 2 mg/dl, creatinine clearance (24 hour collection) >50 cc/min. (Required labs must be within -7 days of catheter placement)
8. Patients must be able to provide written informed consent.
9. Patients with the potential for pregnancy or impregnating their partner must agree to follow acceptable birth control methods to avoid conception. Women of child bearing potential must have negative pregnancy test. The anti-proliferative activity of temsirolimus may be harmful to the developing fetus or nursing infant.
10. Patients must not be allergic to temsirolimus or rapamycin.

Exclusion Criteria:

1. Patients with serious concurrent infection or medical illness, which would jeopardize the ability of the patient to receive the chemotherapy outlined in this protocol with reasonable safety.
2. Patients who are pregnant or breast-feeding.
3. Patients without MRI or CT evidence of measurable, contrast-enhancing residual disease are not eligible.
4. Patients receiving concurrent chemotherapeutic or investigational agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-07; Primary Completion 2010-05; Study Completion 2010-05

PRIMARY OUTCOMES:
Microdialysate torisel concentration | 24 hours

SECONDARY OUTCOMES:
Toxicity assessment | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Olson, MD, Principal Investigator — Emory University Winship Cancer Institute
Locations (1):
- Emory University Winship Cancer Institute, Atlanta, Georgia, United States